CLINICAL TRIAL: NCT04341298
Title: Clinical Evaluation of Avulux® Lenses as an Aid in Reducing the Impact of Migraine Headaches
Brief Title: Use of the Avulux® Lenses as an Aid in Reducing the Impact of Migraine Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avulux, Inc. (Industry)
Collaborators: Imarc Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20200480
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: A minimum of 68 subjects will be randomized in to one of two treatment groups in a one-to-one ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In this study, the investigative Avulux® device shall consist of a pair of optical filters in the form of spectacle lenses, provided in a standard spectacle frame; the lenses contain a dye that effectively blocks light at specified wavelength ranges while minimizing distortion of the visible spectrum. The optical filters block a portion of the optical spectrum that is suspected to stimulate photophobic responses that trigger some, and exacerbate most, migraines.
  The control/sham device for this study shall be a pair of plastic lenses provided in a standard spectacle frame, which will have negligible light-blocking properties at the optical wavelengths which are blocked by the Avulux® device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avulux® device (Experimental): Subjects will be instructed to use the glasses for four weeks. They will be instructed to put the glasses on at the first signs or symptoms consistent with the onset of a migraine attack or at the first onset of aura and keep the glasses on until their headache has resolved.
  Interventions: Other: 11-point pain scale; Other: Headache diary; Device: Avulux®
- Control/sham device (Sham Comparator): Subjects will be instructed to use the glasses for four weeks. They will be instructed to put the glasses on at the first signs or symptoms consistent with the onset of a migraine attack or at the first onset of aura and keep the glasses on until their headache has resolved.
  Interventions: Other: 11-point pain scale; Other: Headache diary; Device: Sham Avulux®

INTERVENTIONS:
Other: 11-point pain scale — Subjects will be asked to rate their headache pain using an 11-point scale, i.e. on an integer scale from 0 to 10 inclusive, with 0 indicating no pain and 10 indicating the worst pain imaginable.
Other: Headache diary — Subjects will be asked to record specific information for the first (and all subsequent) severe or very severe migraine headaches that they experience while enrolled in the study.
Device: Avulux® — Avulux® device
  Arms: Avulux® device
Device: Sham Avulux® — Sham Avulux®
  Arms: Control/sham device

SUMMARY:
The purpose of this research is to assess how well the Avulux® migraine lenses work in reducing the impact of migraine headaches as measured by improvement in an 11-point pain scale after two and four hours of device application, when compared to a control device.

DETAILED DESCRIPTION:
Avulux® is intended to reduce the severity of headache pain in adult patients diagnosed with episodic migraine headaches. In this study, the investigative Avulux® device shall consist of a pair of optical filters in the form of spectacle lenses, provided in a standard spectacle frame; the lenses contain a dye that effectively blocks light at specified wavelength ranges while minimizing distortion of the visible spectrum. The optical filters block a portion of the optical spectrum that is suspected to stimulate photophobic responses that trigger some, and exacerbate most, migraines.

The control/sham device for this study shall be a pair of plastic lenses provided in a standard spectacle frame, which will have negligible light-blocking properties at the optical wavelengths which are blocked by the Avulux® device.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Subject is willing and able to provide written informed consent
* Diagnosis of migraine, based on a history of at least 5 attacks per month with the following primary headache characteristics:

  * Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
  * Headache has at least two of the following characteristics:

    * unilateral location
    * pulsating quality
    * moderate or severe pain intensity
    * aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs)
  * Headache occurs with at least one of the following symptoms:

    * nausea and/or vomiting
    * photophobia and phonophobia
* Subject has experienced at least 4 migraine attacks in the last month, with at least two migraine attacks resulting in severe pain prior to the use of any abortive medications
* Migraines are not attributed to another disorder

Exclusion Criteria:

* Subjects participating in another prospective, interventional clinical study
* Subjects with other light sensitive conditions, such as iritis
* Subjects who have less than 4 headache days per month with the above characteristics
* Chronic migraine subjects (defined as subjects who experience a minimum of 15 headache days per month)
* Subjects with headaches due to medication overuse (defined as regular use of headache medication for a minimum of 10 days per month, for a minimum period of 3 months)
* Subjects who have had any change in their migraine treatment within 4 weeks prior to study enrollment
* Subjects whose family members are currently participating in this study, or are employees of the study site, Avulux, or the coordinating CRO

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Endocrinology Research Associates, Inc., Columbus, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Posternack C, Kupchak P, Capriolo AI, Katz BJ. Targeting the intrinsically photosensitive retinal ganglion cell to reduce headache pain and light sensitivity in migraine: A randomized double-blind trial. J Clin Neurosci. 2023 Jul;113:22-31. doi: 10.1016/j.jocn.2023.04.015. Epub 2023 May 5. PMID 37150129

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avulux® Device | Control/Sham Device
Started | 38 | 40
Completed | 38 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avulux® Device | Control/Sham Device | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (13.3) | 44.3 (13.9) | 46.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 34 | 65
  Black or African-American | 4 | 3 | 7
  Hispanic or Latino | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change in 11-point Pain Scale Score After Two Hours (First Severe Headache)
Description: Change in migraine pain from baseline to 2 hours after device application, based on first severe or very severe migraine headache experienced by a study subject (i.e. baseline pain score of 6 or higher). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: from baseline to 2 hours after device application
Population: The analysis population consists of the participants who experienced a minimum of one severe headache during the study and for whom pain scores were reported at baseline and 2 hours after device application for their first severe headache.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 26 | 29
score on a scale | -1.42 (1.90) | -1.14 (1.43)
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in 11-point Pain Scale Score After Four Hours (First Severe Headache)
Description: Change in migraine pain from baseline to 4 hours after device application, based on first severe or very severe migraine headache experienced by a study subject (i.e. baseline pain score of 6 or higher). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: from baseline to four hours after device application
Population: The analysis population consists of the participants who experienced a minimum of one severe headache during the study and for whom pain scores were reported at baseline and 4 hours after device application for their first severe headache.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 21 | 25
score on a scale | -2.67 (2.67) | -2.80 (2.66)
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Test type: Superiority; p = 0.87, t-test, 2 sided

3. Other Pre Specified Outcome: Number of Subjects With Quantifiable Improvement in Pain Score After Two Hours (First Severe Headache)
Description: Number of subjects who show quantifiable improvement in overall migraine impact, as measured by a change in migraine pain from severe (i.e. baseline pain score of 6 or higher) to mild/no pain (defined as a pain score of 3 or less) after an elapsed time of 2 hours following application of the device, based on first severe or very severe migraine headache experienced by a study subject. Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: from baseline to 2 hours after device application
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 26 | 29
Participants | 2 | 4
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Each subject was stratified by baseline pain score for the first severe headache that they experienced (score of 6-7 vs. 8-10). The total number of subjects, and the number of subjects with a pain score of 3 or less after 2 hours, were tabulated within each stratum. A Cochran-Mantel-Haenszel test was conducted to test the hypothesis of lack of association between the proportion of subjects reporting mild or no symptoms after 2 hours and the type of device, across all strata; Test type: Superiority; p = 0.66, Mantel Haenszel; Subjects were stratified based on baseline pain score (6-7 vs. 8-10) prior to analysis using Cochran-Mantel-Haenszel test

4. Other Pre Specified Outcome: Number of Subjects Who Require the Use of Abortive Medications (First Severe Headache)
Description: Number of subjects who require abortive headache medication (e.g. analgesic or triptan) to control their first severe or very severe migraine headache (i.e. baseline pain score of 6 or higher) within 8 hours following application of the device. Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: baseline to 8 hours after device application
Population: The analysis population consists of the participants who experienced a minimum of one severe headache during the study and who recorded whether abortive medications were used within 8 hours of device application for their first severe headache.
Measure: Count of Participants; unit: Participants
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 26 | 30
Participants | 11 | 11
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Each subject was stratified by baseline pain score for the first severe headache that they experienced (score of 6-7 vs. 8-10). The total number of subjects, and the number of subjects requiring abortive medication within 8 hours were tabulated within each stratum. A Cochran-Mantel-Haenszel test was conducted to test the hypothesis of lack of association between the proportion of subjects requiring abortive medication within 8 hours and the type of device, across all strata; Test type: Superiority; p = 0.59, Mantel Haenszel; [statistical method as in outcome 3, analysis 1]

5. Other Pre Specified Outcome: Number of Subjects Suffering From Light Sensitivity After 2 Hours (First Severe Headache)
Description: Number of subjects suffering from light sensitivity after elapsed time of 2 hours following application of the device, based on first severe or very severe migraine headache experienced by a study subject (i.e. baseline pain score of 6 or higher). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: 2 hours after device application
Population: The analysis population consists of the participants who experienced a minimum of one severe headache during the study and who recorded whether light sensitivity was experienced two hours after device application for their first severe headache.
Measure: Count of Participants; unit: Participants
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 25 | 29
Participants | 9 | 16
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Each subject was stratified by baseline pain score for the first severe headache that they experienced (score of 6-7 vs. 8-10). The total number of subjects, and the number of subjects experiencing light sensitivity after 2 hours, were tabulated within each stratum. A Cochran-Mantel-Haenszel test was conducted to test the hypothesis of lack of association between the proportion of subjects reporting light sensitivity after 2 hours and the type of device, across all strata; Test type: Superiority; p = 0.19, Mantel Haenszel; [statistical method as in outcome 3, analysis 1]

6. Other Pre Specified Outcome: Number of Subjects Suffering From Light Sensitivity After 4 Hours (First Severe Headache)
Description: Number of subjects suffering from light sensitivity after elapsed time of 4 hours following application of the device, based on first severe or very severe migraine headache experienced by a study subject (i.e. baseline pain score of 6 or higher). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: 4 hours after device application
Population: The analysis population consists of the participants who experienced a minimum of one severe headache during the study and who recorded whether light sensitivity was experienced four hours after device application for their first severe headache.
Measure: Count of Participants; unit: Participants
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 20 | 25
Participants | 7 | 10
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Each subject was stratified by baseline pain score for the first severe headache that they experienced (score of 6-7 vs. 8-10). The total number of subjects, and the number of subjects experiencing light sensitivity after 4 hours, were tabulated within each stratum. A Cochran-Mantel-Haenszel test was conducted to test the hypothesis of lack of association between the proportion of subjects reporting light sensitivity after 4 hours and the type of device, across all strata; Test type: Superiority; p = 1.0, Mantel Haenszel; [statistical method as in outcome 3, analysis 1]

7. Post Hoc Outcome: Change in 11-point Pain Scale Score After Two Hours (All Headaches)
Description: Change in migraine pain from baseline to 2 hours after device application, based on all migraine headaches experienced by a study subjects (i.e. baseline pain score of 2 or greater). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: from baseline to 2 hours after device application
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Avulux® Device: Subjects will be instructed to use the glasses for four weeks. They will be instructed to put the glasses on at the first signs or symptoms consistent with the onset of a migraine attack or at the first onset of aura and keep the glasses on until their headache has resolved.
  11-point pain scale: Subjects will be asked to rate their headache pain using an 11-point scale, i.e. on an integer scale from 0 to 10 inclusive, with 0 indicating no pain and 10 indicating the worst pain imaginable.
  Headache diary: Subjects will be asked to record specific information for all migraine headaches (baseline pain score of 2 or greater) that they experience while enrolled in the study.
  Avulux®: Avulux® device
- Control/Sham Device: Subjects will be instructed to use the glasses for four weeks. They will be instructed to put the glasses on at the first signs or symptoms consistent with the onset of a migraine attack or at the first onset of aura and keep the glasses on until their headache has resolved.
  11-point pain scale: Subjects will be asked to rate their headache pain using an 11-point scale, i.e. on an integer scale from 0 to 10 inclusive, with 0 indicating no pain and 10 indicating the worst pain imaginable.
  Headache diary: Subjects will be asked to record specific information for all migraine headaches (baseline pain score of 2 or greater) that they experience while enrolled in the study.
  Sham Avulux®: Sham Avulux®
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 38 | 40
score on a scale | -1.91 (2.13) | -1.05 (1.82)
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Null hypothesis is that 2 hour difference in pain score is equivalent between study arms, after adjusting for baseline pain score and headache medication use; Test type: Superiority; p = 0.021, Mixed Models Analysis; Pain score difference after 2 hours modeled as a function of study arm, baseline pain score and headache medication use

8. Post Hoc Outcome: Change in 11-point Pain Scale Score After Four Hours (All Headaches)
Description: Change in migraine pain from baseline to 4 hours after device application, based on all migraine headaches experienced by a study subjects (i.e. baseline pain score of 2 or greater). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: from baseline to 4 hours after device application
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 38 | 40
score on a scale | -3.46 (2.87) | -2.10 (2.80)
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Null hypothesis is that 4 hour difference in pain score is equivalent between study arms, after adjusting for baseline pain score and headache medication use; Test type: Superiority; p = 0.019, Mixed Models Analysis; Pain score difference after 4 hours modeled as a function of study arm, baseline pain score and headache medication use

9. Post Hoc Outcome: Number of Headaches With Associated Light Sensitivity After 2 Hours (All Headaches)
Description: Number of headaches with associated light sensitivity after elapsed time of 2 hours following application of the device, based on all migraine headaches experienced by study subjects (i.e. baseline pain score of 2 or higher). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: from baseline to 2 hours after device application
Measure: Number; unit: headaches
Units Other Than Participants: headaches
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 38 | 40
Number analyzed (headaches) | 97 | 102
headaches | 31 | 63
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Test type: Superiority — Null hypothesis is that proportion of headaches with light sensitivity experienced after 2 hours is equivalent between study arms, after adjusting for baseline pain score and headache medication use; p = 0.028, Mixed Models Analysis; Proportion of headaches with light sensitivity after 2 hours modeled as a function of study arm, baseline pain score and headache medication use

10. Post Hoc Outcome: Number of Headaches With Associated Light Sensitivity After 4 Hours (All Headaches)
Description: Number of headaches with associated light sensitivity after elapsed time of 4 hours following application of the device, based on all migraine headaches experienced by study subjects (i.e. baseline pain score of 2 or higher). Pain scale is an 11-point scale, with integer values from 0 (no pain) to 10 (worst pain imaginable) inclusive.
Time Frame: from baseline to 4 hours after device application
Measure: Count of Units; unit: headaches
Units Other Than Participants: headaches
Groups:
- Control/Sham Device: Subjects will be instructed to use the glasses for four weeks. They will be instructed to put the glasses on at the first signs or symptoms consistent with the onset of a migraine attack or at the first onset of aura and keep the glasses on until their headache has resolved.
  11-point pain scale: Subjects will be asked to rate their headache pain using an 11-point scale, i.e. on an integer scale from 0 to 10 inclusive, with 0 indicating no pain and 10 indicating the worst pain imaginable.
  Headache diary: Subjects will be asked to record specific information for all migraine headaches (baseline pain score of 2 of greater) that they experience while enrolled in the study.
  Sham Avulux®: Sham Avulux®
Arm/Group | Avulux® Device | Control/Sham Device
Number analyzed (Participants) | 38 | 40
Number analyzed (headaches) | 84 | 86
headaches | 24 | 34
Statistical Analysis 1: Comparison: Avulux® Device vs Control/Sham Device; Null hypothesis is that proportion of headaches with light sensitivity experienced after 4 hours is equivalent between study arms, after adjusting for baseline pain score and headache medication use; Test type: Superiority; p = 0.46, Mixed Models Analysis; Proportion of headaches with light sensitivity after 4 hours modeled as a function of study arm, baseline pain score and headache medication use

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Avulux® Device | Control/Sham Device
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 1/38 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avulux® Device (N=38) | Control/Sham Device (N=40)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution can independently publish 12 months from completion of the Study. Investigator shall submit the manuscript of any proposed publication to Sponsor at least 30 days before publication, and Sponsor shall have the right to review and comment upon the manuscript in order to protect Sponsor's Confidential Information. Upon Sponsor's request, publication shall be delayed up to 90 additional days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04341298/Prot_SAP_000.pdf